CLINICAL TRIAL: NCT02453334
Title: IRON CLAD: Can Iron Lessen Anemia Due to Cancer and Chemotherapy: A Multi-center, Randomized, Double-blinded, Controlled Study to Investigate the Efficacy and Safety of Injectafer® (Ferric Carboxymaltose Injection) in Adults
Brief Title: Can Iron Lessen Anemia Due to Cancer and Chemotherapy: A Study to Investigate the Efficacy and Safety of Injectafer®
Acronym: IRON CLAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1VIT14039
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Results first posted 2021-05-10 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Cancer and Chemotherapy Related Anemia
MeSH Terms: conditions — Neoplasms | interventions — ferric carboxymaltose; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Injectafer (Experimental): 2 doses of Injectafer at 15mg/kg for a maximum single dose of 750mg given 7 days apart for a total of up to 1500mg.
  Interventions: Drug: Injectafer
- Normal Saline (Placebo Comparator): Normal saline administered as an infusion of no more than 250mL infused over 15 minutes.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Injectafer
  Other Names: ferric carboxymaltose injection
  Arms: Injectafer
Other: Normal Saline
  Arms: Normal Saline

SUMMARY:
Phase III, multicenter, randomized, double-blinded, prospective study with two parallel treatment groups. Patients who present to the hematologist/oncologist and satisfy all inclusion and exclusion criteria will be eligible for participation in this 18-week study.

DETAILED DESCRIPTION:
This is a Phase III, multicenter, randomized, double-blinded, prospective study with two parallel treatment groups. Patients who present to the hematologist/oncologist and satisfy all inclusion and exclusion criteria will be eligible for participation in this 18-week study. Subjects who meet all inclusion criteria and no exclusion criteria, will be randomized into the trial (Group A or B).

ELIGIBILITY:
Inclusion Criteria:

* Subjects (male of female) ≥ 18 years of age able to give informed consent to the study.
* Subjects with non-myeloid malignancies
* Receiving chemotherapy as part of their cancer treatment with at least 4 weeks of treatment remaining.
* Screening visit central laboratory hemoglobin (Hgb) ≤11 g/dL, but ≥8 g/dL.
* Ferritin between 100 and 800 ng/mL and transferrin saturation (TSAT) =<35%
* Subjects must have Eastern Coopertative Oncology Group (ECOG) performance status of 0-2.
* Life expectancy of at least 6 months.
* Demonstrate the ability to understand the requirements of the study, willingness to abide by study restrictions and to return for the required assessments.

Exclusion Criteria:

* Previous participation in a ferric carboxymaltose clinical trial.
* Known hypersensitivity reaction to any component of ferric carboxymaltose.
* Subjects with overt bleeding
* Any anemia treatment within 4 weeks before inclusion (oral iron, IV iron, transfusion, or erythropoiesis-stimulating agents).
* Subjects on erythropoiesis-stimulating agents.
* Requiring dialysis for the treatment of chronic kidney disease.
* Any non-viral infection.
* Known positive hepatitis with evidence of active disease.
* Received an investigational drug within 30 days of screening.
* Alcohol or drug abuse within the past 6 months.
* Hemochromatosis or other iron storage disorders.
* Any other laboratory abnormality, medical condition or psychiatric disorders which in the opinion of the Investigator would put the subject's disease management at risk or may result in the subject being unable to comply with study requirements.
* Pregnant or actively trying to become pregnant (Female subjects who are of childbearing age must have a negative pregnancy test at screening and be practicing an acceptable method of birth control during the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2015-05-23 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Compassionate Care Research Group, Inc., Corona, California
  - Compassionate Care Research Group, Inc., Fountain Valley, California
  - Compassionate Care Research Group, Inc., Riverside, California
  - University Cancer Institute, Boynton Beach, Florida
  - AR Development Solutions, Miami Lakes, Florida
  - Lakes Research, Miami Lakes, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Bond Bond Clinic, P.A., Winter Haven, Florida
  - Joliet Oncology Hematology Associates, Joliet, Illinois
  - MId-Illinois Hematology & Oncology Associates, Ltd., Normal, Illinois
  - OSF Saint Anthony Medical Center for Cancer Care, Rockford, Illinois
  - Horizon Oncology Research, Inc., Lafayette, Indiana
  - Michiana Hematology Oncology, PC, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Ashland-Bellefonte Cancer Center, Ashland, Kentucky
  - Rcca Md, Llc, Bethesda, Maryland
  - Antietam Oncology and Hematology Group, P.C., Hagerstown, Maryland
  - North Mississippi and Oncology Associates, Tupelo, Mississippi
  - The Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Richmond University Medical Center, Staten Island, New York
  - Montefiore Medical Center, The Bronx, New York
  - East Chester Cancer Center, The Bronx, New York
  - Waverly Hematology Oncology, Cary, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Charleston Hematology/Oncology Associates, P.A., Charleston, South Carolina
  - Carolina Blood and Cancer Care, PA, Rock Hill, South Carolina
  - Westchase Clinical Associates, Houston, Texas
  - Bon Secours St. Francis Medical Center, Midlothian, Virginia

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Injectafer: 2 doses of Injectafer at 15mg/kg for a maximum single dose of 750mg given 7 days apart for a total of up to 1500mg.
  Injectafer
- Normal Saline: Normal saline administered as an infusion of no more than 250mL infused over 15 minutes.
  Normal Saline
Period: Overall Study
Arm/Group | Injectafer | Normal Saline
Started | 122 | 122
Completed | 81 | 82
Not Completed | 41 | 40
Not completed — Death | 15 | 13
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 5 | 9
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 17 | 13
Not completed — Other reason | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Injectafer | Normal Saline | Total
Number analyzed (Participants) | 122 | 122 | 244
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (10.02) | 63.1 (9.26) | 63.0 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 69 | 136
  Male | 55 | 53 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 119 | 115 | 234
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 117 | 112 | 229
  Race: Black/African-American | 5 | 8 | 13
  Race: Multiple | 0 | 2 | 2
  Race: American Indian/Alaska Native | 0 | 0 | 0
  Race: Asian | 0 | 0 | 0
  Race: Native Hawaiian/Other Pacific Islander | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 22 | 44
  Georgia | 39 | 38 | 77
  Hungary | 26 | 27 | 53
  Poland | 24 | 24 | 48
  Bulgaria | 11 | 11 | 22
Height [Mean (Standard Deviation); unit: cm] | 166.9 (9.5) | 165.9 (9.6) | 166.4 (9.5)
Iron intolerance [Count of Participants; unit: Participants]
  Yes | 3 | 3 | 6
  No | 119 | 119 | 238
ECOG grade [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group. The ECOG grading is 0=fully active
  1. restricted in physical activity
  2. Capable of all self care unable to carry out activities
  3. Confined more than 50% of waking hours
  4. Completely disabled
  Participants
    0 | 39 | 30 | 69
    1 | 75 | 83 | 158
    2 | 8 | 9 | 17
    3 | 0 | 0 | 0
    4 | 0 | 0 | 0
Cancer stage [Count of Participants; unit: Participants] — Stage 0 = No cancer only abnormal cells Stage 1= Small in one area Stage 2 and 3 = Cancer is larger and grown into nearby tissues. Stage 4 = Spread to other parts of body
  Participants
    0 | 2 | 0 | 2
    1 | 0 | 0 | 0
    2 | 2 | 7 | 9
    3 | 9 | 12 | 21
    4 | 81 | 69 | 150
    Unknown | 28 | 34 | 62

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Decrease in Hemoglobin ≥ 0.5 g/dL From Week 3 to Week 18
Description: The following participants will be considered to have met the primary endpoint:
  * Participants with observed Hgb decrease from baseline between 0.5 g/dL to 1.0 g/dL on two consecutive visits between Weeks 3 and 18.
  * Participants with observed Hgb decrease from baseline ≥1.0 g/dL at one visit.
  * Participants who have a non-study intervention prior to Week 18.
  * Participants who discontinue prior to Week 18 for lack of efficacy or adverse events.
Time Frame: Week 3 to Week 18
Measure: Count of Participants; unit: Participants
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 121 | 118
Participants | 42 | 60
Statistical Analysis 1: Comparison: Injectafer vs Normal Saline; Test type: Other; p = 0.0143, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.30 to 0.87]
Statistical Analysis 2: Comparison: Injectafer vs Normal Saline; Test type: Other; Percentage difference = -15.6, 95% CI 2-sided [-28.01 to -3.10]

2. Secondary Outcome: Change in Hemoglobin From Baseline to Week 18 or to Nonstudy Intervention
Description: Nonstudy Intervention is defined as any of the following:
  * Initiation of erythropoietin for any reason
  * Blood transfusion
  * IV iron
  * Prescribed use of oral iron
Time Frame: Baseline to Week 18
Population: Only subjects who completed the study from the Modified intention to treat (mITT) population.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 119 | 118
g/dL
  Baseline | 9.63 (1.000) | 9.75 (1.008)
  Day 7 Change from Baseline: number analyzed (Participants) | 112 | 112
  Day 7 Change from Baseline | 0.27 (0.901) | 0.01 (0.741)
  Week 2 Change from Baseline: number analyzed (Participants) | 107 | 100
  Week 2 Change from Baseline | 0.53 (1.077) | 0.06 (0.937)
  Week 3 Change from Baseline: number analyzed (Participants) | 98 | 103
  Week 3 Change from Baseline | 0.58 (1.015) | 0.04 (1.028)
  Week 6 Change from Baseline: number analyzed (Participants) | 92 | 92
  Week 6 Change from Baseline | 0.84 (1.264) | 0.07 (1.254)
  Week 9 Change from Baseline: number analyzed (Participants) | 85 | 79
  Week 9 Change from Baseline | 0.85 (1.174) | 0.37 (1.512)
  Week 12 Change from Baseline: number analyzed (Participants) | 76 | 67
  Week 12 Change from Baseline | 1.00 (1.202) | 0.74 (1.274)
  Week 15 Change from Baseline: number analyzed (Participants) | 72 | 65
  Week 15 Change from Baseline | 0.97 (1.394) | 0.79 (1.313)
  Week 18/ET Change from Baseline: number analyzed (Participants) | 69 | 63
  Week 18/ET Change from Baseline | 1.04 (1.718) | 0.87 (1.475)

3. Secondary Outcome: Percentage of Participants With Hemoglobin Increase From Baseline ≥ 1 g/dL at Any Postbaseline Visits Without Receiving a Nonstudy Intervention
Description: Summary of number and percentage(%) of participants with Hgb increase ≥ 1 g/dL increase at any time point in the absence of non-study intervention.
Time Frame: Baseline to Week 18
Population: Only subjects who completed the study from the Modified intention to treat (mITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 119 | 118
Participants | 84 | 64
Statistical Analysis 1: Comparison: Injectafer vs Normal Saline; Test type: Other; p = 0.0097, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.04, 95% CI 2-sided [1.19 to 3.50]
Statistical Analysis 2: Comparison: Injectafer vs Normal Saline; Percentage difference; Test type: Other; Percentage difference = 16.4, 95% CI 2-sided [4.19 to 28.51]

4. Secondary Outcome: Percentage of Participants Who Received Nonstudy Intervention
Description: Intervention is defined as any of the following:
  * Initiation of erythropoietin for any reason
  * Blood transfusion
  * IV iron
  * Prescribed use of oral iron
Time Frame: Baseline to week 18
Population: Only subjects who completed the study from the Modified intention to treat (mITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 119 | 118
Participants | 22 | 25
Statistical Analysis 1: Comparison: Injectafer vs Normal Saline; Test type: Other; Percentage difference = -2.7, 95% CI 2-sided [-12.85 to 7.45]
Statistical Analysis 2: Comparison: Injectafer vs Normal Saline; Placebo group was used as the denominator for odds ratio calculation; Test type: Other; p = 0.5758, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.43 to 1.60]

5. Secondary Outcome: Percentage of Participants With Hemoglobin > 12 g/dL in the Absence of Non-study Intervention
Description: as for outcome 4
Time Frame: Baseline to week 18
Population: Only subjects who completed the study from the Modified intention to treat (mITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 119 | 118
Participants | 31 | 24
Statistical Analysis 1: Comparison: Injectafer vs Normal Saline; Test type: Other; p = 0.2772, Cochran-Mantel-Haenszel — Placebo group was used as the denominator for odds ratio calculation; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.76 to 2.56]
Statistical Analysis 2: Comparison: Injectafer vs Normal Saline; Test type: Other; Percentage difference = 5.7, 95% CI 2-sided [-5.01 to 16.43]

6. Secondary Outcome: Time to Hemoglobin Increase ≥ 1 g/dL in the Absence of Non-study Intervention
Description: Participants who discontinued or completed the study, or received a non-study intervention before having an increased in Hgb ≥ 1 g/dL will be censored at last study visit or time of receiving non-study intervention, respectively
Time Frame: Baseline to Week 18
Population: Only subjects who completed the study from the Modified intention to treat (mITT) population.
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 119 | 118
Days
  Q1, 1st quartile | 15 [15 to 20] | 23 [21 to 43]
  Q2, 2nd quartile or median | 43 [22 to 45] | 85 [64 to 106]
  Q3, 3rd quartile | 106 [69 to NA] — Not applicable because insufficient number of participants with events. | NA [126 to NA] — Not applicable because insufficient number of participants with events.
Statistical Analysis 1: Comparison: Injectafer vs Normal Saline; Test type: Other; p = 0.0011, Log Rank; P-value was estimated using logrank test stratified by country

7. Secondary Outcome: Percentage of Participants Requiring a Blood Transfusion
Description: Summary of the number (percentage) of participants requiring a blood transfusion at any time during the trial.
Time Frame: Baseline to week 18
Population: Only subjects who completed the study from the Modified intention to treat (mITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 119 | 118
Participants | 15 | 14
Statistical Analysis 1: Comparison: Injectafer vs Normal Saline; Test type: Other; Percentage difference = 0.7, 95% CI 2-sided [-7.60 to 9.08]
Statistical Analysis 2: Comparison: Injectafer vs Normal Saline; Test type: Other; p = 0.8924, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.49 to 2.29]

8. Secondary Outcome: Percentage of Participants With a Decrease in Hemoglobin ≥ 0.5 g/dL From Baseline to Each Study Visit
Description: Summary of the number and percentage(%) of participants with Hgb decrease (from baseline) ≥ 0.5 g/dL by visit.
Time Frame: Baseline to Day 7
Population: Only participant with both a baseline and at least one post baseline value at Day 7 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 112 | 112
Participants | 18 | 29
Statistical Analysis 1: Comparison: Injectafer vs Normal Saline; Test type: Other; Percentage difference = -9.8, 95% CI 2-sided [-20.41 to 0.77]
Statistical Analysis 2: Comparison: Injectafer vs Normal Saline; The odds ratio (95% [CI) and P-value of treatment effect is based on Cochran-Mantel-Haenszel (CMH) chi-squared test adjusting for country. Placebo group was used as the denominator for odds ratio calculation; Test type: Other; p = 0.0740, Cochran-Mantel-Haenszel; Placebo group was used as the denominator for odds ratio calculation; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.28 to 1.06]

9. Secondary Outcome: Percentage of Participants With a Decrease in Hemoglobin ≥ 0.5 g/dL From Baseline to Each Study Visit
Description: Summary of the number and percentage(%) of participants with Hgb decrease (from baseline) ≥ 0.5 g/dL by visit.
Time Frame: Baseline to Week 2
Population: Only participant with both a baseline and at least one post baseline value at Week 2 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 107 | 100
Participants | 17 | 28
Statistical Analysis 1: Comparison: Injectafer vs Normal Saline; Test type: Other; Percentage difference = -12.1, 95% CI 2-sided [-23.31 to -0.91]
Statistical Analysis 2: Comparison: Injectafer vs Normal Saline; Test type: Other; p = 0.0446, Cochran-Mantel-Haenszel — The odds ratio (95% [CI) and P-value of treatment effect is based on Cochran-Mantel-Haenszel (CMH) chi-squared test adjusting for country; Placebo group was used as the denominator for odds ratio calculation; Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.26 to 0.99]

10. Secondary Outcome: Percentage of Participants With a Decrease in Hemoglobin ≥ 0.5 g/dL From Baseline to Each Study Visit
Description: Summary of the number and percentage(%) of participants with Hgb decrease (from baseline) ≥ 0.5 g/dL by visit.
Time Frame: Baseline to Week 3
Population: Only participant with both a baseline and at least one post baseline value at Week 3 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 98 | 103
Participants | 12 | 33
Statistical Analysis 1: Comparison: Injectafer vs Normal Saline; Test type: Other; Percentage difference = -19.8, 95% CI 2-sided [-30.90 to -8.69]
Statistical Analysis 2: Comparison: Injectafer vs Normal Saline; Test type: Other; p = 0.0010, Cochran-Mantel-Haenszel — [p-value comment as in outcome 9, analysis 2]; Placebo group was used as the denominator for odds ratio calculation; Odds Ratio (OR) = 0.30, 95% CI 2-sided [0.14 to 0.63]

11. Secondary Outcome: Percentage of Participants With a Decrease in Hemoglobin ≥ 0.5 g/dL From Baseline to Each Study Visit
Description: Summary of the number and percentage(%) of participants with Hgb decrease (from baseline) ≥ 0.5 g/dL by visit.
Time Frame: Baseline to Week 6
Population: Only participant with both a baseline and at least one post baseline value at Week 6 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 92 | 93
Participants | 12 | 32
Statistical Analysis 1: Comparison: Injectafer vs Normal Saline; Test type: Other; Percentage difference = -21.4, 95% CI 2-sided [-33.22 to -9.51]
Statistical Analysis 2: Comparison: Injectafer vs Normal Saline; Test type: Other; p = 0.0009, Cochran-Mantel-Haenszel — [p-value comment as in outcome 9, analysis 2]; Odds Ratio (OR) = 0.29, 95% CI 2-sided [0.13 to 0.61] — Placebo group was used as the denominator for odds ratio calculation

12. Secondary Outcome: Percentage of Participants With a Decrease in Hemoglobin ≥ 0.5 g/dL From Baseline to Each Study Visit
Description: Summary of the number and percentage(%) of participants with Hgb decrease (from baseline) ≥ 0.5 g/dL by visit.
Time Frame: Baseline to Week 9
Population: Only participant with both a baseline and at least one post baseline value at Week 9 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 85 | 79
Participants | 9 | 21
Statistical Analysis 1: Comparison: Injectafer vs Normal Saline; Test type: Other; Percentage difference = -16.0, 95% CI 2-sided [-27.73 to -4.26]
Statistical Analysis 2: Comparison: Injectafer vs Normal Saline; Test type: Other; p = 0.0093, Cochran-Mantel-Haenszel — [p-value comment as in outcome 9, analysis 2]; Odds Ratio (OR) = 0.34, 95% CI 2-sided [0.14 to 0.79] — Placebo group was used as the denominator for odds ratio calculation

13. Secondary Outcome: Percentage of Participants With a Decrease in Hemoglobin ≥ 0.5 g/dL From Baseline to Each Study Visit.
Description: Summary of the number and percentage(%) of participants with Hgb decrease (from baseline) ≥ 0.5 g/dL by visit.
Time Frame: Baseline to Week 12
Population: Only participant with both a baseline and at least one post baseline value at Week 12 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 76 | 67
Participants | 8 | 10
Statistical Analysis 1: Comparison: Injectafer vs Normal Saline; Test type: Other; Percentage difference = -4.4, 95% CI 2-sided [-15.37 to 6.57]
Statistical Analysis 2: Comparison: Injectafer vs Normal Saline; Test type: Other; p = 0.4786, Cochran-Mantel-Haenszel — [p-value comment as in outcome 9, analysis 2]; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.26 to 1.89] — Placebo group was used as the denominator for odds ratio calculation

14. Secondary Outcome: Percentage of Participants With a Decrease in Hemoglobin ≥ 0.5 g/dL From Baseline to Each Study Visit.
Description: Summary of the number and percentage(%) of participants with Hgb decrease (from baseline) ≥ 0.5 g/dL by visit.
Time Frame: Baseline to Week 15
Population: Only participant with both a baseline and at least one post baseline value at Week 15 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 72 | 65
Participants | 8 | 12
Statistical Analysis 1: Comparison: Injectafer vs Normal Saline; Test type: Other; Percentage difference = -7.4, 95% CI 2-sided [-19.25 to 4.55]
Statistical Analysis 2: Comparison: Injectafer vs Normal Saline; Test type: Other; p = 0.2084, Cochran-Mantel-Haenszel — [p-value comment as in outcome 9, analysis 2]; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.20 to 1.43] — Placebo group was used as the denominator for odds ratio calculation

15. Secondary Outcome: Percentage of Participants With a Decrease in Hemoglobin ≥ 0.5 g/dL From Baseline to Each Study Visit
Description: Summary of the number and percentage(%) of participants with Hgb decrease (from baseline) ≥ 0.5 g/dL by visit.
Time Frame: Baseline to Week 18
Population: Only participant with both a baseline and at least one post baseline value at Week 18 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 69 | 63
Participants | 12 | 9
Statistical Analysis 1: Comparison: Injectafer vs Normal Saline; Test type: Other; Percentage difference = 3.1, 95% CI 2-sided [-9.33 to 15.54]
Statistical Analysis 2: Comparison: Injectafer vs Normal Saline; Test type: Other; p = 0.6508, Cochran-Mantel-Haenszel; The odds ratio (95% [CI) and P-value of treatment effect is based on Cochran-Mantel-Haenszel (CMH) chi-squared test adjusting for country; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.48 to 3.24] — Placebo group was used as the denominator for odds ratio calculation

16. Secondary Outcome: Time to a Decrease in Hemoglobin ≥ 0.5 g/dL From Baseline to Week 18
Description: Patients who discontinued or completed the study, or received a nonstudy intervention before having an increase in Hgb ≥ 0.5 g/dL were censored at last study visit or time of receiving nonstudy intervention, respectively.
Time Frame: Baseline to Week 18
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 119 | 118
Days
  Q1 | 15 [14 to 43] | 14 [8 to 15]
  Q2 | 127 [106 to NA] — Not available because of the insufficient number of participants with events. | 43 [22 to 64]

17. Secondary Outcome: Time to a Decrease in Hemoglobin ≥ 0.5 g/dL From Baseline to Week 18
Description: as for outcome 16
Time Frame: From Baseline to Week 18
Population: Only subjects who completed the study from the Modified intention to treat (mITT) population.
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 119 | 118
Days
  Q1,1st quartile | 15 [14 to 43] | 14 [8 to 15]
  2nd quartile or median | 127 [106 to NA] — Not available because insufficient number of participants with events. | 43 [22 to 64]
  Q3, 3rd quartile | NA [NA to NA] — Not available because insufficient number of participants with events. | NA [128 to NA] — Not available because insufficient number of participants with events.
Statistical Analysis 1: Comparison: Injectafer vs Normal Saline; Test type: Other; p = 0.0063, Log Rank — P-value was estimated using logrank test stratified by pooled sites

18. Secondary Outcome: Correlation of Change in Hemoglobin With Baseline Hepcidin Level
Description: For participants who receive non-study intervention or early withdraw from the study, the time of intervention or early withdrawal will be considered as end of study, respectively.
Time Frame: Baseline to Week 18.
Population: Only subjects who completed the study from the Modified intention to treat (mITT) population.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 119 | 118
g/dL
  Hepcidin in 1st Tertile | 0.88 (1.892) | 1.13 (1.203)
  hepcidin in 3rd Tertile | 1.28 (1.552) | 0.02 (1.394)

19. Secondary Outcome: Total Score of the Functional Assessment of Chronic Illness Therapy Fatigue(FACIT-Fatigue) Scale Mean Change From Baseline to Week 18
Description: Summary of the actual value and change from baseline in total score of Functional Assessment of Chronic Illness Therapy Fatigue Scale (FACIT-Fatigue Scale). Ranges from 0-52 and higher scores mean better Quality of Life (QOL). Data collected after receiving non-study intervention will not be included in the summary.
Time Frame: Baseline to Week 18
Population: Only subjects who completed the study from the Modified intention to treat (mITT) population.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 119 | 118
Score on a scale
  Baseline: number analyzed (Participants) | 118 | 118
  Baseline | 21.8 (9.47) | 21.5 (8.64)
  Day 7 Change from Baseline: number analyzed (Participants) | 117 | 118
  Day 7 Change from Baseline | -0.8 (6.78) | -0.7 (6.21)
  Week 2 Change from Baseline: number analyzed (Participants) | 110 | 108
  Week 2 Change from Baseline | -0.3 (7.34) | 0.2 (8.13)
  Week 3 Change from Baseline: number analyzed (Participants) | 102 | 108
  Week 3 Change from Baseline | -0.3 (7.75) | -0.6 (7.41)
  Week 6 Change from Baseline: number analyzed (Participants) | 93 | 94
  Week 6 Change from Baseline | -0.2 (9.70) | -0.7 (8.13)
  Week 9 Change from Baseline: number analyzed (Participants) | 87 | 83
  Week 9 Change from Baseline | -0.7 (8.35) | 0.3 (8.22)
  Week 12 Change from Baseline: number analyzed (Participants) | 77 | 73
  Week 12 Change from Baseline | -0.1 (9.82) | -0.5 (8.09)
  Week 15 Change from Baseline: number analyzed (Participants) | 75 | 70
  Week 15 Change from Baseline | -0.1 (9.65) | 0.8 (9.11)
  Week 18 Change from Baseline: number analyzed (Participants) | 72 | 64
  Week 18 Change from Baseline | -1.5 (8.78) | 0.0 (8.92)

ADVERSE EVENTS:
Time Frame: 1 year, 7 months
Arm/Group | Injectafer | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/118
Serious Adverse Events (participants affected / at risk) | 28/121 | 22/118
Other Adverse Events (participants affected / at risk) | 96/121 | 95/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Injectafer (N=121) | Normal Saline (N=118)
Gastrointestinal Disorders (Gastrointestinal disorders) | 7 (7) | 0 (0)
Disease progression (General disorders) | 4 (4) | 4 (4)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 1 (1)
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Blood And Lymphatic System Disorders (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Infections And Infestations (Infections and infestations) | 4 (4) | 3 (3)
Renal And Urinary Disorders (Renal and urinary disorders) | 3 (3) | 2 (2)
Cardiac Disorders (Cardiac disorders) | 2 (2) | 3 (3)
Hepatobiliary Disorders (Hepatobiliary disorders) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Injectafer (N=121) | Normal Saline (N=118)
Diarrhoea (Gastrointestinal disorders) | 15 (15) | 8 (8)
Nausea (Gastrointestinal disorders) | 11 (11) | 11 (11)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 3 (3)
Constipation (Gastrointestinal disorders) | 7 (7) | 3 (3)
Fatigue (General disorders) | 18 (18) | 17 (17)
Asthenia (General disorders) | 10 (10) | 11 (11)
Pyrexia (General disorders) | 6 (6) | 11 (11)
Neutrophil count decreased (Investigations) | 8 (8) | 4 (4)
Platelet count decreased (Investigations) | 8 (8) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 4 (4)
Gamma-glutamyltransferase increased (Injury, poisoning and procedural complications) | 6 (6) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 21 (21) | 14 (14)
Leukopenia (Blood and lymphatic system disorders) | 15 (15) | 13 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (10) | 10 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 19 (19) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 7 (7)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 10 (10)
Infections and Infestations (Infections and infestations) | 16 (16) | 14 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 17 (17)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (7)
Vascular Disorders (Vascular disorders) | 11 (11) | 8 (8)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 2 (2)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 6 (6)
Hepatobiliary Disorders (Hepatobiliary disorders) | 4 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT02453334/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/34/NCT02453334/SAP_001.pdf